CLINICAL TRIAL: NCT03928054
Title: Immediate Effects Of Alliance Therapy In Modulation Of Pain And Disability In Subjects With Knee Osteoarthritis: A Randomized Clinical Trial
Brief Title: Immediate Effects Of Alliance Therapy In Modulation Of Pain And Disability In Subjects With Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculdade de Ciências Médicas da Santa Casa de São Paulo (Other)
Responsible Party: Principal Investigator, Claudio Cazarini Junior, Principal Investigator, Faculdade de Ciências Médicas da Santa Casa de São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Robson Massi
Record Dates: First submitted 2019-04-23; First posted 2019-04-25 (Actual); Last update posted 2019-04-25 (Actual); Status verified 2019-01

CONDITIONS: Arthritis; Knee Osteoarthritis
MeSH Terms: conditions — Arthritis; Osteoarthritis, Knee | interventions — Therapeutic Alliance

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1 "Kinesio Taping® KT" (Experimental): Kinesio Taping® KT
  Interventions: Other: Kinesio Taping and therapeutic alliance
- " Kinesio Taping® with therapeutic alliance KT+AT" (Experimental): Kinesio Taping® with therapeutic alliance
  Interventions: Other: Kinesio Taping and therapeutic alliance

INTERVENTIONS:
Other: Kinesio Taping and therapeutic alliance — bandage used in the treatment of orthopedic diseases and the technique of therapeutic approach in the known patient with therapeutic alliance

SUMMARY:
INTRODUCTION: The Osteoarthritis (OA) is the most common type of joint disease, its features include joint space narrowing, osteophytes formation of the joint margins, motor deficit, reduced strength, and persistent pain. As a treatment option physiotherapy has several resources for the patient approach. However, the effect of treatment is not only the application of therapeutic techniques and resources but also to existing contextual factors such as the therapeutic alliance. OBJECTIVE: To assess the effects of an intervention with the focus on positive therapeutic alliance in subjects OA knee on pain and disability. METHODS: This is a randomized study of two arms with a blind evaluator. 40 subjects were randomized into 2 groups: group 1 "Kinesio Taping® KT" group 2 " Kinesio Taping® with therapeutic alliance KT+AT". Both groups received the application of Kinesio Taping® method as the concepts of the original method. The group "KT+AT" session was conducted in order to increase the relationship between the therapist and the patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients with both sexes from 40 to 80 years old
* who underwent imaging examination evidencing grade II or III knee osteoarthritis according to the Kellgren and Lawrence classification
* who were referred to the physiotherapy service by a physician.

Exclusion Criteria:

* Patients who are unable to walk
* with a history of cancer
* associated neurological diseases
* morbid obesity

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2016-01-01 (Actual); Study Completion 2016-07-01 (Actual)

PRIMARY OUTCOMES:
Pain intensity: VAS | 12 weeks
  Pain intensity was assessed using a visual analogic scale (VAS) of 11 items (0 to 10) (22), in which the patient measured the intensity of pain, with 0 = "no pain" and 10 = "worst possible pain

CONTACTS AND LOCATIONS:
Locations (1):
- Claudio Cazarini Júnior, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lawrence RC, Felson DT, Helmick CG, Arnold LM, Choi H, Deyo RA, Gabriel S, Hirsch R, Hochberg MC, Hunder GG, Jordan JM, Katz JN, Kremers HM, Wolfe F; National Arthritis Data Workgroup. Estimates of the prevalence of arthritis and other rheumatic conditions in the United States. Part II. Arthritis Rheum. 2008 Jan;58(1):26-35. doi: 10.1002/art.23176. PMID 18163497